CLINICAL TRIAL: NCT00865995
Title: Pepsin as a Biomarker for Aspiration Due to Gastroesophageal Reflux
Brief Title: Pepsin As A Biomarker For Aspiration
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Nikki Johnston, Assistant Professor, Medical College of Wisconsin
Other Study IDs: CHW 08/26; GC 636
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-10

CONDITIONS: Aspiration; Gastroesophageal Reflux
Keywords: pepsin; aspiration; GE reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tracheal fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: patients undergoing elective procedures with intubation and no known respiratory pathology
  Interventions: Procedure: Tracheal Lavage
- 2: patients with tracheostomy
- 3: patients with chronic lung disease or respiratory symptoms undergoing bronchoscopy

INTERVENTIONS:
Procedure: Tracheal Lavage — Tracheal Lavage will be performed on the control population patients and the tracheal fluid obtained from this procedure will be used as the research sample.
  Groups: 1

SUMMARY:
Evaluation of tracheal pepsin as a biomarker for aspiration

DETAILED DESCRIPTION:
Aspiration is well recognized in children who have chronic lung disease or who are intubated. There is a known association between gastroesophageal reflux (GER) and aspiration. The distinction between aspiration of swallowed material, such as food and the aspiration of refluxed gastric contents is important. Determining whether an aspiration syndrome in an individual is due to GER may be difficult. The most widely used test to determine whether GER is the cause of aspiration involves staining bronchoalveolar lavage (BAL) fluid for lipid laden macrophages (LLM) based on the hypothesis that refluxed and aspirated fluid is phagocytosed by tracheal macrophages.

Pepsinogen is a protein unique to gastric chief cells and also requires acidic conditions for activation. Therefore the presence of pepsin in BAL fluid should only be found when gastric fluid is aspirated. In previous studies, pepsin has been detected in the tracheal fluid of children with chronic lung disease. Thus far, studies of this material have been small, not all have control groups, and LLM were not looked for in all studies.

Based on previous studies and the need to improve diagnostic methods, the following aims are proposed:

1. to determine the frequency of pepsin contamination of children without chronic respiratory disease undergoing elective surgery with intubation
2. to determine frequency of tracheal pepsin and lipid laden macrophages (LLM) in children with chronic respiratory disease or symptoms and in children with tracheostomies
3. to compare the presence or absence and concentration of pepsin to the presence of LLM
4. to relate the presence or absence and concentration of pepsin to clinical status To achieve these aims, BAL fluid will be obtained from subject patients and controls. These fluids will be transported to the research lab and stored on ice until analysis. Determination of LLM will be done in children undergoing diagnostic bronchoscopy in the clinical lab of CHW per routine. BAL analysis will consist of Western blot staining for the presence of pepsin. Demographic data will also be collected from the medical record.

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria of study population

Exclusion Criteria:

* Lack of informed consent/assent
* Pulmonary disease in normal controls

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Normal children undergoing general endotracheal anesthesia Children with tracheostomies Children undergoing bronchoscopy Intubated children in PICU
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2008-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
pepsin concentration | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Nikki Johnston, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States